CLINICAL TRIAL: NCT00005460
Title: Predictors of Cardiovascular Disease in the Elderly
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4904; R01HL044689 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2000-05

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Cerebrovascular Accident; Coronary Disease; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction; Stroke; Coronary Disease; Hypertension

SUMMARY:
To evaluate factors associated with cardiovascular morbidity and mortality in a cohort of 795 men and women aged 75 years or older at the time of a comprehensive examination conducted between 1984 and 1987.

DETAILED DESCRIPTION:
BACKGROUND:

The study was needed because evidence in 1991 suggested that cardiovascular risk factors which had been identified by studies of middle-aged populations did not have the same predictive value in the elderly; especially the "oldest old" aged 75 and above.

DESIGN NARRATIVE:

The study analyzed data that had been collected over the years. At the time of the analysis, mortality follow-up was complete for over 99 percent of subjects, and incident morbidity information was available for myocardial infarction, coronary bypass surgery and stroke. The database included measurements which allowed: 1) prospective analyses of the effects of putative cardiovascular risk factors on disease incidence in the elderly, 2) prospective analyses of the impact of change in risk factors on events in the elderly, 3) exploration of risk factors not classically associated with cardiovascular events in younger populations but which may be important in the very old, and, 4) cross-sectional description of putative risk factors in an aged population.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-01; Study Completion 1992-12 (Actual)

REFERENCES:
- [Background] Langer RD, Criqui MH, Barrett-Connor EL, Klauber MR, Ganiats TG. Blood pressure change and survival after age 75. Hypertension. 1993 Oct;22(4):551-9. doi: 10.1161/01.hyp.22.4.551. PMID 8406660